CLINICAL TRIAL: NCT00617552
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Assess Efficacy and Safety of TZP-101 When Administered as 30 Minute i.v. Infusion for POI to Subjects Undergoing Major Open Abdominal Surgery
Brief Title: Safety and Efficacy of IV Infusion of TZP-101 for POI After Major Open Abdominal Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tranzyme, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TZP-101-CL-P005
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Postoperative Ileus
Keywords: postoperative ileus; POI; major open abdominal surgery
MeSH Terms: interventions — Glucose; Water; ulimorelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 1 (Placebo Comparator)
  Interventions: Drug: 5% dextrose in water
- 2 (Experimental)
  Interventions: Drug: TZP-101
- 3 (Experimental)
  Interventions: Drug: TZP-101
- 4 (Experimental)
  Interventions: Drug: TZP-101
- 5 (Experimental)
  Interventions: Drug: TZP-101
- 6 (Experimental)
  Interventions: Drug: TZP-101
- 7 (Experimental)
  Interventions: Drug: TZP-101
- 8 (Experimental)
  Interventions: Drug: TZP-101

INTERVENTIONS:
Drug: 5% dextrose in water — 60 ml IV infusion over 30 minutes
  Other Names: D5W
  Arms: 1
Drug: TZP-101 — 20 micrograms/kg IV 2ml/minute for 30 minutes
  Arms: 2
Drug: TZP-101 — 40 micrograms/kg IV 2 ml/minute for 30 minutes
  Arms: 3
Drug: TZP-101 — 80 micrograms/kg IV 2ml/minute for 30 minutes
  Arms: 4
Drug: TZP-101 — 160 micrograms/kg IV 2ml/minute over 30 minutes
  Arms: 5
Drug: TZP-101 — 320 micrograms/kg IV 2ml/minute for 30 minutes
  Arms: 6
Drug: TZP-101 — 480 micrograms/kg IV 2ml/minute over 30 minutes
  Arms: 7
Drug: TZP-101 — 600 micrograms/kg IV 2ml/minute for 30 minutes
  Arms: 8

SUMMARY:
The purpose of this study is to determine whether TZP-101 is effective in the management of post operative ileus in subjects undergoing major open abdominal surgery (i.e. partial large bowel resection).

DETAILED DESCRIPTION:
Subjects will be randomized according to an adaptive randomization procedure.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following inclusion criteria may be enrolled in the study:

* Male or Female, 18 to 80 years of age, inclusive
* If female, post-menopausal for the past 12 months, surgically sterile (i.e. tubal ligation, hysterectomy), or using an adequate method of birth control (i.e., oral contraceptives, double barrier method, IUD cover or sterilized partner
* Subject is scheduled to undergo a partial large bowel resection with primary anastomosis - See Appendix II
* Subject's body weight is ≤100kg
* Subject is scheduled to receive postoperative pain management with i.v. opioids
* Subject is scheduled to have nasogastric tube removed at the end of surgery
* Subject is scheduled to be offered liquids on postoperative day 1
* Subject is scheduled to be encouraged for ambulation on postoperative day 1
* Subject is scheduled to be offered solid food on postoperative day 2

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria may not be enrolled in the study:

* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450(men)/ >470(women) milliseconds)
* Subject has history of additional risk factors for Torsades de Pointes (heart failure, hypokalemia, family history of Long QT Syndrome)
* Subject requires use of concomitant medication that prolongs the QT interval - List provided in Study Procedures Manual
* Subject requires use of concomitant medication that is a known to interact with isoenzyme CYP3A4
* Subject has complete bowel obstruction
* Subject is scheduled to receive a thoracic epidural
* Subject is scheduled to receive total colectomy, colostomy, or ileostomy
* Subject is scheduled to receive a lower anterior resection
* Subject is scheduled for laparoscopic procedure
* Subject is scheduled to receive prophylactic antiemetics post surgery; however subjects may receive intraoperatively as part of the anesthesia protocol and postoperative antiemetics for symptomatic treatment
* Subject has significant impairment of liver or renal function (ALT/AST 2 ½ times the upper limit of normal; creatinine clearance < 50mL/min.)
* Subject has a psychiatric disorder or cognitive impairment that would interfere with participation in the study
* Subject has severe cardiovascular, pulmonary, hematological diseases
* Subject has participated in an investigational study 30 days prior or received TZP-101 90 days prior to the study initiation
* Subject is pregnant (confirmed by quantitative serum pregnancy test) or is breast-feeding
* Subject has a known history of Hep B, Hep C or HIV
* Subject has a known history of drug or alcohol abuse
* Subject has a recent, adult history of clinically significant hypersensitivity reaction(s) to any drug

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Time to recovery of gastrointestinal function as defined by the time to first bowel movement. | 7 days of dosing plus 7 days after administration of last dose

SECONDARY OUTCOMES:
time to tolerance of first solid food | 7 days post administration of last dose

CONTACTS AND LOCATIONS:
Locations (27):
- United States (10):
  - Office of Dr. Phillip Fleshner, Los Angeles, California
  - University of Miami Clinic, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Northwestern University, Chicago, Illinois
  - Univ. of Maryland, R.A. Cowley Shock Trauma Center, Baltimore, Maryland
  - Baystate Medical Center/Baystate Health, Springfield, Massachusetts
  - Michigan State/Spectrum Health, Grand Rapids, Michigan
  - Stony Brook University Hospital, Stony Brook, New York
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - The Methodist Hospital, Houston, Texas
- India (8):
  - St. John's Hospital, Bangalore, Karnataka
  - Stanley Medical College, Chennai
  - Asian Institute of Gastroenterology, Hyderabad
  - Nizams Institute of Medical Science, Hyderabad
  - Mediciti Hospitals, Hyderabad
  - Amrita Institute of Medical Sciences, Kochi
  - Lakeshore Hospital, Kochi
  - Sanjay Gandhi Post-Graduate Institute of Medical Sciences, Lucknow
- Romania (9):
  - Clinica de Chirugie General IV, Spitalul Universitar, Bucharest
  - Clinica de Chirugie Generala I, Spitalul Universitar, Bucharest
  - Clinica de Chirugie Generala III, Spitalul Universitar, Bucharest
  - Institul Clinic Fundeni, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Spitalul Clinic Coltea, Bucharest
  - Spitalul Clinic de Urgenta Floreasca, Bucharest
  - Spitalul Urg. SF. Pantelimon, Bucharest
  - Spitalul Universitar Elias, Bucharest